CLINICAL TRIAL: NCT03448627
Title: Physiological Responses to Maximal Exercise Capacity and Muscle Strength in Survived Hematopoietic Stem Cell Transplantation Recipients
Brief Title: Physical Impairments in Allogeneic-HSCT
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: GaziUniversity6
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Stem Cell Transplantation
Keywords: stem cell transplantation; Pulmonary Functions; muscle strength; exercise capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: HSCT recipients: Pulmonary functions [spirometry], maximal exercise capacity [Modified-Incremental Shuttle Walk Test (ISWT)], inspiratory and expiratory muscle strength (MIP and MEP, respectively) [mouth pressure device] and peripheral muscle strength [hand-held dynamometer] were evaluated in allogeneic HSCT recipients (n=66).Vital signs, dyspnea and fatigue perception [Modified Borg Scale] were recorded as pre-post measurements of Modified-ISWT.
- Group 2: healthy individuals: Healthy individuals (n=50) were selected from individuals without known and diagnosed any chronic diseases. Similar measurements were applicated in healthy individuals.

SUMMARY:
Pulmonary functions, exercise capacity and muscle strength deteriorate in survived hematopoietic stem cell transplantation (HSCT) recipients due to toxic effects of chemotherapy, radiotherapy, conditioning regimens and/or corticosteroid use before HSCT, prolonged stay of recipients in rooms with laminar airflow and strict infection control rules during process of HSCT. There are also limited numbers of studies demonstrated pulmonary function abnormalities, decreased maximal exercise capacity, respiratory and peripheral muscle weakness in recipients. Current study was planned since no study compared pulmonary functions, maximal exercise capacity, respiratory and peripheral muscle strength between recipients and healthy individuals in the literature.

DETAILED DESCRIPTION:
Treatments of hematologic malignancies consist of chemotherapy, radiotherapy, surgery, medical treatment, supportive care and/or hematopoietic stem cell transplantation (HSCT) which is resulted in early or late adverse effects on body systems, tissues and organs. Physical deconditioning is also observed in patients with hematologic malignancies because of reasons such as neurotoxic and pulmonary toxic effects of long term these anticancer treatments, immobilization, recommendation of resting and avoiding intense exercise, nutrition problems, severe anemia and thrombocytopenia etc. For these reasons, normal physical activities may not be kept on by patients which induces decreased physical performance.

The HSCT provides longer survival with standard treatments for patients with hematological malignancies while it increases risk of HSCT-related toxicity, complications and even mortality. Infectious and non-infectious pulmonary complications occur in about 60% of HSCT recipients and intensive-care unit support is also required in one-third of recipients for these reasons. Restrictive lung disease prior to allogeneic HSCT is related to early respiratory failure, non-relapse mortality and respiratory muscle weakness in post transplantation period. Therefore pulmonary restriction is considered as a risk factor for complications or failure of HSCT. Moreover it is known that carbon monoxide diffusing capacity of lungs which is the most common abnormality seen in pulmonary function test, respiratory muscle strength and functional exercise capacity are reduced in the majority of patients before HSCT. In addition to muscle weakness and decreased exercise capacity at prior to HSCT, patients experience more reduction in both inspiratory and expiratory muscles and exercise capacity after HSCT. Unfortunately, exercise capacity and peripheral muscle strength are decreased in HSCT recipients in spite of doing regular and planned exercise during acute process of HSCT. The average reduction in functional exercise capacity of recipients is 48 m. As shown in the literature, limited number of study has used evaluation of maximal exercise capacity with Modified-Incremental Shuttle Walk Test (ISWT) in HSCT patients and recipients. On the other hand, it has been reported that ISWT is a reliable test and has no adverse event or side effects for HSCT recipients in these studies, as well. Despite the fact that there is no negative feedback related to using of this test in recipients, no study comprehensively demonstrated influence of HSCT on maximal exercise capacity.

Impairments in pulmonary functions, respiratory muscle strength and maximal exercise capacity have been demonstrated in limited number of studies. Moreover, there is no study compared pulmonary functions, respiratory muscle strength and maximal exercise capacity between HSCT recipients and healthy individuals. Therefore investigators aimed to compare aforementioned outcomes between recipients and healthy individuals.

ELIGIBILITY:
Inclusion Criteria for recipients:

* between ages of 18 and 70
* under standard medical treatment
* underwent allogeneic HSCT who were at minimum 100 days status post-transplantation

Exclusion Criteria for recipients:

* having cognitive disorder, orthopedic or neurological disease with a potential to affect assessment of maximal exercise capacity,
* having comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute respiratory or other infections,
* having problems like visual and mucositis which may prevent measurements,
* acute hemorrhage anywhere in the body,
* hemoglobin value less than 8 g/L and platelet count less than 10.000 mm3

Inclusion Criteria for healthy individuals:

* being individuals without known and diagnosed any chronic diseases
* not actively smoking
* their cigarette exposure is not greater than 5 pack*year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 66 recipients underwent allogeneic HSCT who were at minimum 100 days status post-transplantation compared with 50 healthy individuals.
  All recipients transplanted at the Bone Marrow Transplantation Unit of University Faculty of Medicine. All measurements were done by a physiotherapist at Cardiopulmonary Unit of University Faculty of Health Science Department of Physiotherapy and Rehabilitation. Demographic and clinical characteristics of all participants were recorded. Study was planned as retrospective, cross sectional and approved by the local Ethics Committee. Informed consent was obtained from all individual participants included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Modified-Incremental Shuttle Walk Test (ISWT) | 15-20 minutes
  This test was used to evaluate maximal exercise capacity

SECONDARY OUTCOMES:
pulmonary function test | 5 minutes
  This test was evaluated using a spirometry
inspiratory and expiratory muscle strength (MIP, MEP) | 5-10 minutes
  Respiratory muscle strength was evaluated with a mouth pressure device
Quadriceps femoris muscle strength | 5 minutes
  Peripheral muscle strength was evaluated with a hand-held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Gülsan Türköz Sucak, Principal Investigator — Bahçeşehir University
Locations (1):
- Gazi University Faculty of Health Science Department of PhysioTherapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Result] Kovalszki A, Schumaker GL, Klein A, Terrin N, White AC. Reduced respiratory and skeletal muscle strength in survivors of sibling or unrelated donor hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):965-9. doi: 10.1038/bmt.2008.15. Epub 2008 Feb 11. PMID 18264142
- [Result] Morishita S, Kaida K, Yamauchi S, Sota K, Ishii S, Ikegame K, Kodama N, Ogawa H, Domen K. Relationship between corticosteroid dose and declines in physical function among allogeneic hematopoietic stem cell transplantation patients. Support Care Cancer. 2013 Aug;21(8):2161-9. doi: 10.1007/s00520-013-1778-7. Epub 2013 Mar 9. PMID 23475197
- [Result] Knols RH, de Bruin ED, Uebelhart D, Aufdemkampe G, Schanz U, Stenner-Liewen F, Hitz F, Taverna C, Aaronson NK. Effects of an outpatient physical exercise program on hematopoietic stem-cell transplantation recipients: a randomized clinical trial. Bone Marrow Transplant. 2011 Sep;46(9):1245-55. doi: 10.1038/bmt.2010.288. Epub 2010 Dec 6. PMID 21132025
- [Result] Shelton ML, Lee JQ, Morris GS, Massey PR, Kendall DG, Munsell MF, Anderson KO, Simmonds MJ, Giralt SA. A randomized control trial of a supervised versus a self-directed exercise program for allogeneic stem cell transplant patients. Psychooncology. 2009 Apr;18(4):353-9. doi: 10.1002/pon.1505. PMID 19117328
- [Result] Morishita S, Kaida K, Yamauchi S, Wakasugi T, Ikegame K, Ogawa H, Domen K. Relationship of physical activity with physical function and health-related quality of life in patients having undergone allogeneic haematopoietic stem-cell transplantation. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12669. Epub 2017 Feb 21. PMID 28220548
- [Result] Bargi G, Guclu MB, Aribas Z, Aki SZ, Sucak GT. Inspiratory muscle training in allogeneic hematopoietic stem cell transplantation recipients: a randomized controlled trial. Support Care Cancer. 2016 Feb;24(2):647-659. doi: 10.1007/s00520-015-2825-3. Epub 2015 Jul 2. PMID 26135532
- [Result] Bird L, Arthur A, Niblock T, Stone R, Watson L, Cox K. Rehabilitation programme after stem cell transplantation: randomized controlled trial. J Adv Nurs. 2010 Mar;66(3):607-15. doi: 10.1111/j.1365-2648.2009.05232.x. PMID 20423395